CLINICAL TRIAL: NCT00438152
Title: A 24-week, Randomized, Open-label, 2-arm Study to Compare the Safety, Efficacy and Tolerability of Invirase® Tablets With Ritonavir Versus Kaletra® Tablets in HIV 1 Infected Adults on a Kaletra® Based Regimen With 2 Nucleosides/Nucleotides
Brief Title: Lopinavir Capsules to Kaletra or Invirase Tablets
Acronym: LoCKIT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Royal Free Hampstead NHS Trust (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Dr. Mike Youle, Royal Free Hampstead NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MV20507
Record Dates: First submitted 2007-02-19; First posted 2007-02-21 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2007-02

CONDITIONS: HIV Infections
Keywords: Lopinavir; Saquinavir; Lipids; HIV-1; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Saquinavir; Lopinavir; Ritonavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Invirase® tablets (Active Comparator)
  Interventions: Drug: Saquinavir (Invirase®)
- Kaletra® tablets (Active Comparator)
  Interventions: Drug: Lopinavir/ritonavir (Kaletra®)

INTERVENTIONS:
Drug: Saquinavir (Invirase®) — Saquinavir 1000mg + Ritonavir 100mg Bd for 24 weeks
  Other Names: Invirase®
  Arms: Invirase® tablets
Drug: Lopinavir/ritonavir (Kaletra®) — Lopinavir/ritonavir 400/100 mg BD 24 weeks
  Other Names: Kaletra®
  Arms: Kaletra® tablets

SUMMARY:
This study will compare the benefit for patients switching from Kaletra® to Invirase® tablets over remaining on Kaletra® (based on randomization), to elicit the lipid benefits inferred in previous studies

DETAILED DESCRIPTION:
This is a prospective, phase IV, multicentre, randomised, open-label, 2-arm, 24-week study. Approximately 130 HIV-1 infected patients on a stable antiretroviral regimen containing Kaletra® with 2 nucleoside/nucleotide analogues will be randomized to 1 of 2 treatment arms: saquinavir with ritonavir 1000/100 mg BID (using Invirase® tablets) or lopinavir/ritonavir 400/100 mg BID (using Kaletra® tablets).Eligibility for enrollment will be determined at a screening visit that will occur within 30 days of the baseline visit. Protocol-defined study assessments will take place at clinic visits at the end of Weeks 4, 12, and 24.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-nursing females >18 years of age
* Seropositive for HIV-1
* On an antiretroviral combination of Kaletra® with 2 nucleoside/nucleotide analogues for at least 6 months
* HIV-1 RNA viral load <50 copies/mL (2 consecutive measurements in the prior 6 months) plus screening viral load <50 copies/ml.
* Ability and willingness to provide written informed consent and adhere to the study regimen
* Females of childbearing potential must have a documented negative serum or urine pregnancy test at screening/baseline and ensure that 2 reliable forms of contraception are being used, including a barrier method, for the duration of the study and for 90 days after the last dose of study medication

Exclusion Criteria:

* Documented virological failure on a protease inhibitor ARV regimen prior to commencing Kaletra® regimen
* Documented protease mutation (one or more from the following list) prior to commencing Kaletra® regimen:
* M46I/L/V, I47A/V, G48V/M, I50V, F53L/Y, I54L/M/V/A/T/S, V82A/T/S/F/M/L, I84A/V/C, L90M
* Patients with acute hepatitis B or C infection
* Females who are pregnant, breast-feeding, or who plan to become pregnant or breast-feed during the study·
* Significant renal dysfunction (creatinine clearance [CrCl] <60 mL/min) and/or hepatic impairment (aspartate aminotransferase/alanine aminotransferase [AST/ALT] >3 X ULN and/or documented liver cirrhosis)

Note: The site will calculate each patient's CrCl using the Cockcroft-Gault formula [28] as shown below:

CrCl = [140 - age (yr)] × weight (kg) × constant 72 × serum creatinine (Cr) (mg/dL) where, constant = 1 for men and 0.85 for women

* Any current known clinical or laboratory parameter of ACTG Grade 4 (see Appendix 4). However, asymptomatic Grade 4 abnormalities will be permitted at the discretion of the investigator if deemed clinically appropriate. Abnormalities deemed insignificant by the investigator must be discussed with the sponsor prior to enrollment.
* Evidence of active, untreated opportunistic infection, intercurrent illness, drug toxicity or any other condition such that in the judgment of the investigator the patient would not be able to take or continue a prescribed antiretroviral regimen
* Malignancy requiring chemotherapy or radiotherapy
* Known hypersensitivity to any of the prescribed antiretroviral drugs or formulation components
* Evidence of alcohol and/or drug or substance abuse that in the judgment of the investigator would likely result in the patient being unreliable in fulfilling the conditions of the protocol
* History of psychological illness or conditions that in the judgment of the investigator might interfere with the patient's ability to understand the requirements of the study
* History of drug non-adherence that in the judgment of the investigator would result in the patient being unreliable in fulfilling the conditions of this protocol
* Patients who had received an investigational new drug within the last 4 weeks
* Currently taking, or anticipate taking during the course of the study, any drug contraindicated with the antiretroviral drugs they have been randomized to receive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2006-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the lipid benefits of Invirase® tablets with ritonavir versus Kaletra® tablets in HIV-1 infected adults on an antiretroviral regimen containing Kaletra® with two nucleosides/nucleotides | 24 weeks

SECONDARY OUTCOMES:
To evaluate the efficacy of Invirase® tablets with ritonavir versus Kaletra® tablets in HIV-1 infected adults on an ARV regimen containing Kaletra® with 2 nucleosides/nucleotides. | 4 weeks, 12 weeks and 24 weeks.
To evaluate additional safety and tolerability of Invirase® tablets with ritonavir versus Kaletra® tablets in HIV-1 infected adults on an antiretroviral regimen containing Kaletra® with 2 nucleosides/nucleotides. | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Mike S Youle, MD MB ChB, Principal Investigator — Royal Free Hampstead NHS Trust
Locations (1):
- Royal Free Hampstead NHS Trust, London, United Kingdom